CLINICAL TRIAL: NCT03835078
Title: Performance of Aspheric Hydrogel Lenses After a Refit With Sphere Silicone Hydrogel Lenses for 4 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EX-MKTG-98
Record Dates: First submitted 2019-01-31; First posted 2019-02-08 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Masking Description: Study lenses will be transferred, by an assistant, out of their packaging to unmarked new contact lens cases filled with unpreserved sterile saline just prior to dispensing to maintain subject masking of the study lenses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- methalfilcon A contact lenses / fanfilcon A contact lenses (Experimental): All subjects will first wear methafilcon A contact lenses for four (4) weeks of daily wear, then be refitted with fanfilcon A toric contact lenses for four (4) weeks of daily wear.
  Interventions: Device: methafilcon A contact lenses; Device: fanfilcon A contact lenses

INTERVENTIONS:
Device: methafilcon A contact lenses — Bilateral daily wear of methafilcon A contact lenses
Device: fanfilcon A contact lenses — Bilateral daily wear of fanfilcon A contact lenses

SUMMARY:
The aim of this prospective study is to evaluate the clinical performance of habitual wearers of methafilcon A aspheric lenses after a refit with fanfilcon A sphere lenses for 4 weeks of daily wear.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft contact lens wearer
* Has a contact lens spherical prescription between - 0.25 to - 8.00 (inclusive)
* Have no less than -0.75D (Diopter) of astigmatism in both eyes
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter
* Patient contact lens refraction should fit within the available parameters of the study lenses
* Is willing to comply with the wear schedule (at least 5 days per week, >8 hours/day assuming there are no contraindications for doing so)
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has a Contact Lens (CL) prescription outside the range of the available parameters of the study lenses
* Has a spectacle cylinder of ≥ 1.00D (Diopter) in either eye
* Has a history of not achieving comfortable Contact Lens (CL) wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Velazquez, MSc FIACLE, Principal Investigator — School of Optometry, National Autonomous University
Locations (1):
- Optometry Clinic, National Autonomous University, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 subjects were enrolled but three subjects did not satisfy the minimum number of days / hours of wear during the study and excluded from all the analysis.
Period: Overall Study
Arm/Group | Methalfilcon A Contact Lenses / Fanfilcon A Contact Lenses
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Lens Centration Assessment by the Investigator - Methafilcon A Contact Lenses
Description: Lens centration assessment using 3-point scale (1=optimal centration, 2=decentration acceptable, 3=decentration unacceptable).
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Methalfilcon A Contact Lenses: All subjects will wear methafilcon A contact lenses for four (4) weeks of daily wear.
  methafilcon A contact lenses: Bilateral daily wear of methafilcon A contact lenses
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
percentage of participants
  Optimal Centration | 100
  Decentration Acceptable | 0
  Decentartion Unacceptable | 0

2. Primary Outcome: Percentage of Participants With Lens Centration Assessment by the Investigator - Methafilcon A Contact Lenses
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
percentage of participants
  Optimal Centration | 100
  Decentration Acceptable | 0
  Decentration Unacceptable | 0

3. Primary Outcome: Percentage of Participants With Lens Centration Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 1
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Fanfilcon A Contact Lenses: All subjects will wear fanfilcon A toric contact lenses for four (4) weeks of daily wear.
  fanfilcon A contact lenses: Bilateral daily wear of fanfilcon A contact lenses
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
percentage of participants
  Optimal Centration | 100
  Decentration Acceptable | 0
  Decentration Unacceptable | 0

4. Primary Outcome: Percentage of Participants With Lens Centration Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
percentage of participants
  Optimal Centration | 100
  Decentration Acceptable | 0
  Decentration Unacceptable | 0

5. Primary Outcome: Percentage of Participants With Lens Centration Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
percentage of participants
  Optimal Centration | 100
  Decentartion Acceptable | 0
  Decentration Unacceptable | 0

6. Primary Outcome: Percentage of Participants With Corneal Coverage Assessment by the Investigator - Methafilcon A Contact Lenses
Description: Corneal coverage is collected on a YES/NO response. Yes - lens covers the cornea, No - lens does not cover the cornea
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
percentage of participants
  Yes | 97.4
  No | 2.6

7. Primary Outcome: Percentage of Participants With Corneal Coverage Assessment by the Investigator - Methafilcon A Contact Lenses
Description: Corneal coverage is collected on a YES/NO response. Yes - lens covers the cornea, No - lens does not cover the cornea
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
percentage of participants
  Yes | 100
  No | 0

8. Primary Outcome: Percentage of Participants With Corneal Coverage Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: Corneal coverage is collected on a YES/NO response. Yes - lens covers the cornea, No - lens does not cover the cornea
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
percentage of participants
  Yes | 100
  No | 0

9. Primary Outcome: Percentage of Participants With Corneal Coverage Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: Corneal coverage is collected on a YES/NO response. Yes - lens covers the cornea, No - lens does not cover the cornea
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
percentage of participants
  Yes | 100
  No | 0

10. Primary Outcome: Percentage of Participants With Corneal Coverage Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: Corneal coverage is collected on a YES/NO response. Yes - lens covers the cornea, No - lens does not cover the cornea
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
percentage of participants
  Yes | 100
  No | 0

11. Primary Outcome: Post-blink Movement Assessment by the Investigator - Methafilcon A Contact Lenses
Description: Post-blink movement, was rated at each visit using a 0-4 scale (0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 1.90 (0.3)

12. Primary Outcome: Post-blink Movement Assessment by the Investigator - Methafilcon A Contact Lenses
Description: as for outcome 11
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 1.95 (0.3)

13. Primary Outcome: Post-blink Movement Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 11
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 1.97 (0.2)

14. Primary Outcome: Post-blink Movement Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 11
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 1.97 (0.2)

15. Primary Outcome: Post-blink Movement Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 11
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 2.0 (0.2)

16. Primary Outcome: Lens Tightness Assessment by the Investigator - Methafilcon A Contact Lenses
Description: Lens tightness was assessed using the push-up test and a 0 - 100% continuous scale (where 0% =falls from cornea without lid support, 50% = optimum and 100%=no movement).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 53.59 (9.6)

17. Primary Outcome: Lens Tightness Assessment by the Investigator - Methafilcon A Contact Lenses
Description: as for outcome 16
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 52.31 (6.5)

18. Primary Outcome: Lens Tightness Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 16
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 50.38 (1.8)

19. Primary Outcome: Lens Tightness Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 16
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 50.64 (3.3)

20. Primary Outcome: Lens Tightness Assessment by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 16
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 50.51 (3.2)

21. Primary Outcome: Overall Lens Fit Acceptance by the Investigator - Methafilcon A Contact Lenses
Description: Lens fit acceptance was evaluated using a 0 - 4 scale 0=Should not be worn, 1=Borderline but unacceptable, 2=Minimal acceptable, early review, 3=Not perfect but okay to dispense, 4=perfect
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 3.69 (0.6)

22. Primary Outcome: Overall Lens Fit Acceptance by the Investigator - Methafilcon A Contact Lenses
Description: as for outcome 21
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 3.74 (0.5)

23. Primary Outcome: Overall Lens Fit Acceptance by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 21
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 3.97 (0.2)

24. Primary Outcome: Overall Lens Fit Acceptance by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 21
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 3.92 (0.3)

25. Primary Outcome: Overall Lens Fit Acceptance by the Investigator - Fanfilcon A Contact Lenses
Description: as for outcome 21
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
units on a scale | 3.95 (0.3)

26. Secondary Outcome: Average Daily Wearing Time - Methafilcon A Contact Lenses
Description: Average daily wearing time response by the subject
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours / day
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
hours / day | 12.1 (4.0)

27. Secondary Outcome: Average Daily Wearing Time - Fanfilcon A Contact Lenses
Description: Average daily wearing time response by the subject.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours / day
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
hours / day | 12.2 (2.6)

28. Secondary Outcome: Average Daily Wearing Time - Fanfilcon A Contact Lenses
Description: Average daily wearing time response by the subject
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours / day
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
hours / day | 12.3 (2.6)

29. Secondary Outcome: Average Comfortable Wearing Time - Methafilcon A Contact Lenses
Description: Average comfortable wearing time - response by the subject
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours / day
Arm/Group | Methalfilcon A Contact Lenses
Number analyzed (Participants) | 39
hours / day | 10.0 (3.2)

30. Secondary Outcome: Average Comfortable Wearing Time - Fanfilcon A Contact Lenses
Description: Average comfortable wearing time - response by the subject
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours / day
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
hours / day | 9.6 (3.0)

31. Secondary Outcome: Average Comfortable Wearing Time - Fanfilcon A Contact Lenses
Description: Average comfortable wearing time - response by the subject
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours / day
Arm/Group | Fanfilcon A Contact Lenses
Number analyzed (Participants) | 39
hours / day | 9.7 (2.9)

ADVERSE EVENTS:
Time Frame: From baseline up to 8 weeks
Groups:
- Methafilcon A: All subjects will wear methafilcon A contact lenses for four (4) weeks of daily wear, then be refitted with fanfilcon A toric contact lenses for four (4) weeks of daily wear.
  methafilcon A contact lenses: Bilateral daily wear of methafilcon A contact lenses
- Fanfilcon A: All subjects will wear methafilcon A contact lenses for four (4) weeks of daily wear, then be refitted with fanfilcon A toric contact lenses for four (4) weeks of daily wear.
  fanfilcon A contact lenses: Bilateral daily wear of fanfilcon A
Arm/Group | Methafilcon A | Fanfilcon A
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT03835078/Prot_SAP_001.pdf